CLINICAL TRIAL: NCT06983847
Title: Observational Study on Vitamin C-Injektopas® 7.5g in Patients With Vitamin C Deficiency Due to Acute and Chronic Diseases
Brief Title: A Long-term Observational Study to Describe the Use of Vitamin-C Injektopas® 7.5 g in Patients With Vitamin C Deficiency
Status: Recruiting | Type: Observational
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 214A18VCAT
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Deficiency, Vitamin C; Chronic Disease; Acute Disease
MeSH Terms: conditions — Ascorbic Acid Deficiency; Chronic Disease; Acute Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vit C deficiency in acute diseases: Patients with vitamin C deficiency due to a acute underlying disease treated with Vitamin-C injektopas® 7.5 g
- Vit C deficiency in chronic diseases: Patients with vitamin C deficiency due to a chronic underlying disease treated with Vitamin-C injektopas® 7.5 g

SUMMARY:
The goal of this observational study is to learn more about the disease and the symptoms where the product will use and in which patient groups. Further on, it is interesting to know clinical pictures, the symptoms improve. Patients with acute or chronical disease with vitamin c deficiency could be involved.

The main questions it aims to answer are:

* how do the symptoms of the disease change
* how is the tolerability

DETAILED DESCRIPTION:
The aim of this long-term observational study is to document the use of Vitamin C Injektopas® 7.5g in patients with vitamin C deficiency. The deficiency condition can be diagnosed either by laboratory diagnosis or clinically, i.e. symptomatically on the basis of general vitamin C deficiency symptoms (e.g. weakness, fatigue, susceptibility to infections and psychological complaints such as depressive moods) through to more specific deficiency symptoms, which are primarily related to impaired collagen formation and therefore primarily affect connective tissue, blood vessels, cartilage and bones. These include, above all, haemorrhages in the skin, inflamed and bleeding gums - through to tooth loss, joint effusions, pain in the joints, bones and muscles as well as poorly healing wounds, etc.

The survey should be used to assess the disease underlying the vitamin C deficiency (the so-called underlying disease), the reduction in the symptoms of the disease under therapy and also the tolerability. Both acute and chronic underlying diseases should be taken into account.

In addition to the symptom enquiry, the global assessment of the efficacy and tolerability of therapy with Vitamin C Injektopas® 7.5g is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vitamin C deficiency
* Age ≥ 18 years

Exclusion Criteria:

* Hypersensitivity to the active ingredient or any of the excipients
* Oxalate urolithiasis
* Iron storage disease (thalassemia, hemochromatosis, sideroblastic anemia) or recent red blood cell transfusion
* Renal insufficiency
* Glucose-6-phosphate dehydrogenase deficiency/defect
* Pregnant/breastfeeding women

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a vitamin C deficiency due to acute or chronic underlying diseases
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-12 (Actual); Primary Completion 2028-01-12 (Estimated); Study Completion 2028-11-14 (Estimated)

PRIMARY OUTCOMES:
change in general and disease-specific symptoms | therapy duration, an expected average of 3 weeks (for acute diseases) or 12 weeks (for chronic diseases)
  The main aim was to measure the success of the treatment with Vitamin C-Injektopas® 7,5g by the documentation of the change in general and disease-specific symptoms.
  The symptoms are measured by a score:
  0 = not present, 1 = slightly, 2 = moderate and 3 = strong
  The change of the symptoms is measured in change groups:
  * number of patients with improved symptoms
  * number of patients with unchanged symptoms
  * number of patients with worsened symptoms

SECONDARY OUTCOMES:
Global assessment of efficacy of treatment with Vitamin C-Injektopas® 7,5g | therapy duration, an expected average of 3 weeks (for acute diseases) or 12 weeks (for chronic diseases)
  Global assessment of efficacy is measured by a score:
  * Very good efficacy (complete regression of symptoms)
  * Good efficacy (symptoms was much improved)
  * Moderate efficacy (symptoms was slightly improved)
  * No efficacy (symptoms remained unchanged)
  * No efficacy (symptoms worsened)
Dosage scheme | Number of infusions through study completion, up to appr. 12 weeks
  Number of infusions during the observational time
Global Assessment of Tolerability | on last visit, an expected average of 3 weeks (for acute diseases) or 12 weeks (for chronic diseases)
  Global Assessment of Tolerability of the treatment with Vitamin C-Injektopas® 7,5g
  Global assessment of tolerability is measured by a score:
  * Very good tolerability (no side effects)
  * Poor tolerability (side effects occurred)
Quality of life in chronic disease (Numeric Scale) | therapy duration, an expected average of 12 weeks (for chronic diseases)
  Quality of life in chronic disease, Numeric Scale (NRS) from 0 - 10

CONTACTS AND LOCATIONS:
Overall Officials: Holger Michels, Study Director, Study Director — Pascoe Pharmazeutische Praeparate GmbH
Locations (1):
- Multiple Physicians from Austria, Vienna, Etc., Austria, Austria

IPD SHARING:
Plan to Share IPD: No
All data are anonymous. Patient data list only will be sent to regulatory authorities.